CLINICAL TRIAL: NCT07277075
Title: Probiotic Intervention and Its Influence on Serum Leucine-Rich Alpha-2 Glycoprotein 1 Levels in Acne Vulgaris Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Zeinab Ali Awad Menesy, MBBCH of Dermatology, Venereology and Andrology, Benha University, Benha, Egypt., Benha University
Other Study IDs: 40-10-2024
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Probiotic; Influence; Serum Leucine-Rich Alpha-2 Glycoprotein 1; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Participants with clinically diagnosed mild to moderate acne vulgaris (AV) based on the Glycosaminoglycans (GAGs).
  Interventions: Diagnostic Test: Serum Leucine-rich alpha-2 glycoprotein 1 (LRG1) level
- Control group: Apparently healthy controls matched for age and sex
  Interventions: Diagnostic Test: Serum Leucine-rich alpha-2 glycoprotein 1 (LRG1) level

INTERVENTIONS:
Diagnostic Test: Serum Leucine-rich alpha-2 glycoprotein 1 (LRG1) level — Serum Leucine-rich alpha-2 glycoprotein 1 (LRG1) levels were assessed in acne vulgaris participants and healthy controls.

SUMMARY:
This study aimed to assess the serum level of Leucine-rich alpha-2 glycoprotein 1 (LRG1) in Acne vulgaris (AV) individuals and evaluate the effect of probiotic therapy on these serum levels.

DETAILED DESCRIPTION:
Acne vulgaris (AV) is a common inflammatory disorder of the pilosebaceous units, characterized by the presence of inflammatory, non-inflammatory, or a combination of both types of lesions.

Recent attention has turned toward biomarkers that reflect the inflammatory activity in acne and might act as indicators of disease severity, treatment response, or prognostic risk. One such candidate is Leucine-rich alpha-2 glycoprotein 1 (LRG1).

Probiotics are live microorganisms that, when administered in sufficient quantities, can modulate the composition of the gut microbiota, helping reduce microbial dysbiosis, regulate the immune response, and decrease inflammatory mediators, thereby reducing systemic inflammatory burden, which is called the gut-skin-axis relationship.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sexes.
* Had not used systemic or topical acne therapy for at least two months or two weeks before the research, respectively.
* Participants with clinically diagnosed mild to moderate acne vulgaris (AV) based on the Global Acne Grading System (GAGS)

Exclusion Criteria:

* Pregnancy.
* Lactation.
* History of hypersensitivity to probiotic components.
* Smoking.
* Presence of infections.
* Autoimmune or malignant diseases.
* Receiving any systemic therapy likely to affect the microbiome or inflammatory biomarkers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study was conducted on all participants enrolled from the Dermatology & Andrology Outpatient Clinic at Benha University Hospital, Egypt, between October 2024 and September 2025.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Serum Leucine-Rich Alpha-2 Glycoprotein 1 Level | 12 weeks after the therapy
  Serum Leucine-Rich Alpha-2 Glycoprotein 1 Level was assessed.

SECONDARY OUTCOMES:
Acne severity | 12 weeks after the therapy
  Acne severity was assessed based on Global Acne Grading System (GASA) score is considered as 1-18 "mild," 19-30 "moderate," 31-38 "severe," and >39 "very severe"
Patient satisfaction | 12 weeks after the therapy
  Patient satisfaction was evaluated using the Likert scale, with response options ranging from 1 = very dissatisfied to 5 = very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.